CLINICAL TRIAL: NCT02663921
Title: Determination of the Minimal Dose of Visible Light Required to Achieve Immediate Pigment Darkening, Persistent Pigment Darkening, and Delayed Tanning for Fitzpatrick Skin Types IV-VI Utilizing Two Visible Light Sources.
Brief Title: Visible Light Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-02039
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Skin Disease; Pigment Disorders
Keywords: Fitzpatrick Skin-Type; Melanin; Ultraviolet Light (UV)
MeSH Terms: conditions — Skin Diseases; Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): Healthy volunteers without cutaneous disorders associated with pigmentary changes
  Interventions: Other: Part A: Baseline-Week 2; Other: Part B: Week 4-Week 12

INTERVENTIONS:
Other: Part A: Baseline-Week 2 — The study doctor will shine 2 different light bulbs (one a regular or incandescent bulb and the other an LED light bulb) on 12 different areas of patients skin approximately 6 square centimeters in size (less than 1 square inch or the size of your thumb nail). Each light bulb will be exposed to your skin for approximately 20 - 35 minutes. After exposure, the study doctor will perform skin assessments at 3 time points:
  1. Immediately after the light exposure;
  2. 30 minutes after light exposure; and
  3. 1 hour after light exposure.
Other: Part B: Week 4-Week 12 — The study doctor will perform the same 4 skin assessments used in Part A at each visit to assess potential changes in your skin: Digital Photography
  1. Visual Clinical Assessment
  2. Spectroscopy
  3. Colorimetry

SUMMARY:
The purpose of this study is to learn more about the potential effects of visible light on the skin. More specifically, this study will examine whether an incandescent lamp (light bulb) or LED light bulb can cause skin to become darker. Investigators will determine the minimum threshold dose required to achieve immediate pigmentation darkening (IPD), persistent pigmentation darkening (PPD), and delayed tanning (DT) for Fitzpatrick skin types IV - VI utilizing two visible light sources.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy volunteer with Fitzpatrick skin types I-VI;
* Agree to abide by the Investigator's guidelines regarding photosensitizing drugs and photoprotection;
* Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form;
* Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

* Women who are lactating, pregnant, or planning to become pregnant;
* Patients with a recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post-inflammatory hyperpigmentation;
* Patients with a known history of photosensitivity disorders;
* Photosensitizing medications may be continued throughout of the study at the discretion of the investigator ;
* Patients with a known history of melanoma or non-melanoma skin cancers;
* Concomitant use of tanning beds;
* Sun exposure of the irradiated or control areas;
* Patients with serious systemic disease.
* Patients with a known history of hypersensitivity to adhesives including adhesive tape.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Diffuse Reflectance Spectroscopy (DRS) to examine the optical properties of melanin and deoxyhemoglobin | 12 weeks
Quantification of the scattering and absorption properties of the skin in which the beam of light will penetrate using DRS | 12 weeks
Measurement of pigmentation changes induced by the two light sources using diffuse reflectance spectrometer | 12 weeks
Measurement of pigmentation changes induced by the two light sources using Colorimetry | 12 weeks
Measurement of pigmentation changes induced by the two light sources using Cross-Polarized Digital Photography | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Soter, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States